CLINICAL TRIAL: NCT01680783
Title: Mechanical Ventilation in Patients With \Respiratory Failure: A Comparison of Face Mask and Non Invasive Ventilation Via a Helmet Device
Brief Title: Non-Invasive Ventilation Via a Helmet Device for Patients Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-1391
Record Dates: First submitted 2012-08-29; First posted 2012-09-07 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Acute Respiratory Distress Syndrome; Shock; Ventilatory Failure; Cardiogenic Pulmonary Edema
Keywords: noninvasive ventilation; acute hypoxemic respiratory failure; Acute respiratory distress syndrome; shock
MeSH Terms: conditions — Respiratory Distress Syndrome; Shock; Hypoventilation; Respiratory Insufficiency | interventions — Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Other): Patients who require noninvasive ventilation via Face mask for more than 8 hours will continue using noninvasive ventilation via facemask.
  Interventions: Other: Noninvasive ventilation via facemask
- Non invasive ventilation via helmet (Experimental): Patients requiring more than 8 hours of noninvasive ventilation via facemask will switch to non-invasive ventilation using a helmet instead of face mask for treatment of respiratory failure
  Interventions: Device: Non invasive ventilation using a helmet hyperbaric device

INTERVENTIONS:
Device: Non invasive ventilation using a helmet hyperbaric device — Patients randomized to the intervention group will receive noninvasive ventilation delivered via a latex-free helmet connected to the ventilator by conventional tubing.
  If endotracheal intubation is required, the helmet will be removed and the patient will be intubated without delay.
  Other Names: Sea-Long medical treatment hood
  Arms: Non invasive ventilation via helmet
Other: Noninvasive ventilation via facemask — Patients assigned to the conventional ventilation group will continue noninvasive ventilation via facemask
  Other Names: mechanical ventilation
  Arms: Usual Care

SUMMARY:
The objective of our study is to evaluate the efficacy of helmet ventilation as compared with Face mask in patients with respiratory failure.

DETAILED DESCRIPTION:
Respiratory failure is often treated with endotracheal intubation and mechanical ventilation. Although, the institution of mechanical ventilation is considered life saving, the associated complications of tracheal stenosis, ventilator associated pneumonia, barotrauma , and neuromuscular weakness are not without considerable morbidity and mortality.

Non-invasive ventilation has demonstrated significant benefit in patients with hypercapnic respiratory failure from COPD, acute cardiogenic pulmonary edema, and hypoxemic respiratory failure in immunocompromised patients.

Despite the advantages of non-invasive ventilation via facemask, some patients fail because of mask intolerance and severity of disease. Further limitation to facemask non-invasive ventilation is that the seal integrity is lost when higher pressures are required. Unfortunately, certain types of respiratory failure such as that due to hypoxemia or shock may require such higher pressures.

In an attempt to improve patient tolerability and deliver higher pressures, a transparent helmet has been proposed as a novel interface for non-invasive ventilation. It encloses the entire head and neck of the patient. The design of the helmet confers some important advantages: 1) the transparency allows the patient to interact with the environment; 2) the lack of contact to the face lowers the risk of skin necrosis; 3) the helmet avoids problems of leaking with higher airway pressures that are seen with the face mask; 4) it can be applied to any patient regardless of facial contour.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years of age who require noninvasive ventilation via facemask for >8hours
* Intact airway protective gag reflex
* Able to follow instructions

Exclusion Criteria:

* Cardiopulmonary arrest
* Glasgow coma scale <8
* Absence of airway protective gag reflex
* Elevated intracranial pressure
* Tracheostomy
* Upper airway obstruction
* Pregnancy.
* Patients who refuse to undergo endotracheal intubation, whatever the initial therapeutic approach

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Kress, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Patel BK, Wolfe KS, Pohlman AS, Hall JB, Kress JP. Effect of Noninvasive Ventilation Delivered by Helmet vs Face Mask on the Rate of Endotracheal Intubation in Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2016 Jun 14;315(22):2435-41. doi: 10.1001/jama.2016.6338. PMID 27179847

RESULTS

PARTICIPANT FLOW:
Groups:
- Non Invasive Ventilation Via Helmet: Patients requiring more than 8 hours of noninvasive ventilation via facemask will switch to non-invasive ventilation using a helmet instead of face mask for treatment of respiratory failure
  Non invasive ventilation using a helmet hyperbaric device: Patients randomized to the intervention group will receive noninvasive ventilation delivered via a latex-free helmet connected to the ventilator by conventional tubing.
  If endotracheal intubation is required, the helmet will be removed and the patient will be intubated without delay.
Period: Overall Study
Arm/Group | Usual Care | Non Invasive Ventilation Via Helmet
Started | 39 | 44
Completed | 39 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Non Invasive Ventilation Via Helmet | Total
Number analyzed (Participants) | 39 | 44 | 83
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60.9 [56.4 to 71.1] | 58 [49.8 to 67.8] | 59 [52 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 21 | 24 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 28 | 50
  White | 16 | 14 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Need for Endotracheal Intubation
Description: Number of patients requiring endotracheal intubation after application of helmet device
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Non Invasive Ventilation Via Helmet
Number analyzed (Participants) | 39 | 44
Participants | 24 | 8

2. Secondary Outcome: Hospital Length of Stay
Description: Days spent in hospital at time of enrollment
Time Frame: Duration of hospital stay
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Usual Care | Non Invasive Ventilation Via Helmet
Number analyzed (Participants) | 39 | 44
days | 15.2 [7.8 to 19.7] | 10.1 [6.5 to 15.9]

3. Secondary Outcome: Number of Participants Functional Status After Discharge
Description: Telephone survey of patients 1, 6, and 12 months after discharge to assess need for re-hospitalization, admission to nursing home, and functional status (ability to complete ADLs and IADLs independently)
Time Frame: Measured at 1, 6, and 12 months after hospital discharge (to span time frame of up to 80 weeks depending on length of hospitalization)
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Non Invasive Ventilation Via Helmet
Number analyzed (Participants) | 39 | 44
Participants | 6 | 22

4. Secondary Outcome: Ventilator-free Days
Description: Duration of mechanical ventilation via endotracheal tube
Time Frame: number of days in the hospital
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Usual Care | Non Invasive Ventilation Via Helmet
Number analyzed (Participants) | 39 | 44
days | 12.5 [0.49 to 28] | 28 [13.7 to 28]

5. Secondary Outcome: Hospital Mortality
Description: Death from any cause during hospitalization at time of enrollment
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Non Invasive Ventilation Via Helmet
Number analyzed (Participants) | 39 | 44
Participants | 19 | 12

6. Secondary Outcome: Intensive Care Unit Length of Stay
Description: Number of days admitted to a medical intensive care unit
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Usual Care | Non Invasive Ventilation Via Helmet
Number analyzed (Participants) | 39 | 44
days | 7.8 [3.9 to 13.8] | 4.7 [2.5 to 8.7]

7. Other Pre Specified Outcome: ICU Complications
Description: ICU complications will include rates of Ventilator associated pneumonia, Barotrauma, Gastrointestinal hemorrhage, Pulmonary embolism, Sacral Decubitus ulcer, Delirium, ICU acquired weakness
Time Frame: 6 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Readmission to the Intensive Care Unit
Description: Measure the need for readmission to the intensive care unit during initial hospitalization at time of enrollment
Time Frame: 6 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Discharge Location
Description: Measure the location (ie home, rehabilitation center, nursing home) that patients are discharged to
Time Frame: 6 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Improvement of Oxygenation
Description: Improvement of oxygenation-defined as PaO2/FiO2 ≥ 200 or increase from baseline by 100
Time Frame: 2 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Usual Care | Non Invasive Ventilation Via Helmet
All-Cause Mortality (participants affected / at risk) | 22/39 | 12/44
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/44
Other Adverse Events (participants affected / at risk) | 0/39 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No